CLINICAL TRIAL: NCT02019615
Title: Repeated tDCS in Chronic Minimally Conscious State Patients : a Sham-controlled Randomized Double Blind Study
Brief Title: tDCS in MCS: Repeated Stimulations
Acronym: tDCS in MCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Aurore Thibaut, MSc, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009/201/B
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Patients in Minimally Conscious State After a Severe Brain Injury (e.g., Anoxia, Traumatic Brain Injury, Stroke)
Keywords: disorders of consciousness; minimally conscious state; traumatic brain injury; stroke; transcranial direct current stimulation
MeSH Terms: conditions — Hypoxia; Brain Injuries, Traumatic; Stroke; Consciousness Disorders; Persistent Vegetative State | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anodal stimulation (Active Comparator): Patients received anodal tDCS (on the left dorsolateral prefrontal cortex) every day for 5 days (tDCS of 2mA during 20minutes). A CRS-R is performed at baseline (before the first stimulation) and after each tDCS. A final CRS-R is performed one week after the end of the session to assess the potential long term effects of the tDCS.
  Interventions: Device: transcranial direct current stimulation
- sham stimulation (Sham Comparator): Patients received sham tDCS (5 secondes of stimulation) every day for 5 days. A CRS-R is performed at baseline (before the first stimulation) and after each tDCS. A final CRS-R is performed one week after the end of the session.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — anodal transcranial direct current stimulation on the left dorsolateral prefrontal cortex for the anodal session and sham stimulation (5secondes of tDCS) for the sham session

SUMMARY:
In this study researchers will apply transcranial direct current stimulation (tDCS) for 5 consecutive days in chronic patients in minimally conscious state (MCS).

2 sessions of 5 days of stimulation will be realized, one anodal and one sham. After each stimulation, behavioral improvement will be assessed with the Coma Recovery Scale Revised (CRS-R). A final assessment will be done one week after the end of the sessions to assess the long term effect of the tDCS.

DETAILED DESCRIPTION:
Positive effects of tDCS in patients in MCS was showed in a recent study published in Neurology. But the effects went down after 1 or 2 hours. To increase the lasting of the effects, a new study will evaluate the effects of tDCS on the left prefrontal dorsolateral cortex for 5 consecutive days in chronic patients in MCS.

2 sessions of 5 days of stimulation will be realized, one session will be real (anodal stimulation) and one placebo (sham stimulation). After each stimulation, behavioral improvement will be assessed with the Coma Recovery Scale Revised (CRS-R). A final assessment will be done one week after the end of the sessions to assess the long term effect of the tDCS.

Researchers expected to see an improvement of the CRS-r total score at the end of the anodal session and that this improvement persists for a week.

ELIGIBILITY:
Inclusion Criteria:

* post comatose patients
* patients in minimally conscious state
* patients with stable condition
* patients free of sedative drugs and Na+ or Ca++ blockers (e.g., carbamazepine) or NMDA receptor antagonist (e.g., dextromethorphan)

Exclusion Criteria:

* premorbid neurology antecedent
* patients in coma or vegetative state
* patients < 3 months after the acute brain injury
* patients with a metallic cerebral implant or a pacemaker (in line with the safety criteria for tDCS in humans)

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in the CRS-R total score | after each stimulation and one week later for anodal and sham sessions (total: 1 month)
  Improvement of the CRS-R total score after the end of the anodal session and one week later but no change for the sham session.

SECONDARY OUTCOMES:
Influence of the time since insult | one month
  Influence of the time since insult of the results. We expected that the longer a patient is in MCS, the lower is his/her improvement after the tDCS session.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liège, Liège, Liège, Belgium